CLINICAL TRIAL: NCT01213615
Title: Hancock II Ultra Porcine Bioprosthesis Hemodynamic Study
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Other Study IDs: Rev B February 4, 2010
Record Dates: First submitted 2010-07-26; First posted 2010-10-04 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Aortic Heart Valve Diseases
MeSH Terms: interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- all patients eligible for implantation of a Hancock II Ultra
  Interventions: Device: Valve replacement

INTERVENTIONS:
Device: Valve replacement — Aortic valve replacement of Hancock II Ultra porcine bioprosthesis

SUMMARY:
Since the first implant in September 1982, the Medtronic Hancock® II has provided more than 20 years of excellent hemodynamic performance and durability. Design improvements over the past generations include: low profile, flexible stent, Supra-X™ supra-annular placement, T6 anti-calcification tissue treatment, modified fixation process, CINCH® advanced implant system and ULTRA™ minimized sewing ring. Valve sizing is a critical consideration in obtaining optimal hemodynamic performance. This is particular true in small aortic roots. A critical issue is the size of the prosthesis in relation to the patient's annulus.

The objective of this clinical study is to evaluate, at six and twelve months, the hemodynamic performance of the HancockÒ Ultra™ bioprosthesis in the aortic position, to analyze the incidence of patient prosthesis mismatch, correlation of gradients, and to ascertain frequency at which a larger valve size is used vs. a patient's debrided annulus diameter.

ELIGIBILITY:
Inclusion Criteria:

* Patients who require aortic valve replacement with or without coronary artery bypass grafting or surgical treatment of atrial fibrillation or mitral valve repair.
* Patients who are able to provide informed consent.

Exclusion Criteria:

* Concomitant procedures other than coronary artery bypass grafting, surgical treatment of atrial fibrillation or mitral valve repair.
* Patients indicated for receiving a mechanical prosthesis.
* Patients who will have a replacement of existing valve prosthesis.
* Patients refusing or not able to provide informed consent.
* Patients requiring emergency surgery.
* Patients unable to participate in follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population includes all patients who require aortic valve replacement for heart valve disease (acquired or congenital) and who are candidates for a bioprosthetic valve. Patients will be informed about the aspects of this study and will be asked to give their Informed Consent.
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2008-08; Primary Completion 2013-10 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is the hemodynamic performance of the bioprosthesis at 6 and 12 months after surgery. | 6 and 12 months after surgery
  This will be measured by comparing the mean aortic valve gradients pre- and post-surgery.Left ventricular mass regression will be compared pre operative and at 6 months follow-up. The follow-up data at 12 months will be used to see if there was any improvement with the 6 months follow-up visit. .

SECONDARY OUTCOMES:
The secondary objective of the study is the incidence of patient prosthesis mismatch (PPM). | 5 to 15 days post procedure
  This is measured by collecting valve sizing data during implant and the ultimate valve sizes used for implant

CONTACTS AND LOCATIONS:
Locations (5):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Italy (2):
  - Azienda Ospedaliera Sant'Anna e San Sebastiano, Caserta
  - Azienda Universitaria S. Maria della Misericordia, Udine
- Leiden University Medical Center, Leiden, Netherlands
- The Cardiothoracic Centre Liverpool NHS Trust, Liverpool, United Kingdom